CLINICAL TRIAL: NCT07010380
Title: A Multicenter Prospective Paired Observational Study Evaluating the Performance of the PTFinder Dual-Channel Near-Infrared and White-Light Imaging System With AI-Assisted Analysis for Rapid Identification of Parathyroid Glands in Surgical Specimens
Brief Title: Dual-Channel Near-Infrared Autofluorescence Imaging and AI Analysis to Locate Parathyroid Glands (PTFinder)
Acronym: PTFinder
Status: Recruiting | Type: Observational
Sponsor: Bo Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Bo Wang,MD, Director, Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: PTFinder 3 Dual
Record Dates: First submitted 2025-06-01; First posted 2025-06-08 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Neoplasms; Hyperparathyroidism; Parathyroid Gland
Keywords: Near-Infrared Autofluorescence (NIRAF); Parathyroid Identification; PTFinder Device; Dual-Channel Imaging; Rapid PTH Test Strip; Thyroidectomy Specimen; Ex-Vivo Fluorescence Camera; Sensitivity and Specificity; Artificial Intelligence; Deep Learning; Computer Vision; NIRAF 3 Dual; PTFinder 3 Dual; PTFinder 3.0 Dual; NIRAF 3.0 Dual
MeSH Terms: conditions — Thyroid Neoplasms; Hyperparathyroidism; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Surgical Specimen Cohort: Adults (≥18 y) undergoing thyroid or parathyroid surgery; their excised specimens will be imaged ex vivo with the PTFinder device for parathyroid-gland identification.
  Interventions: Device: PTFinder Dual-Channel NIR Autofluorescence Imaging System; Other: Offline Machine-Learning Algorithm (PTFinder-AI Beta)

INTERVENTIONS:
Device: PTFinder Dual-Channel NIR Autofluorescence Imaging System — Ex vivo, non-contact imaging of resected thyroid/parathyroid specimens; captures near-infrared autofluorescence and overlays it on white-light video to highlight parathyroid glands (2-5 min per specimen).
Other: Offline Machine-Learning Algorithm (PTFinder-AI Beta) — training/validation on de-identified NIR/RGB frames.

SUMMARY:
This study tests PTFinder, a dual-camera system that makes parathyroid glands glow on screen by capturing their natural near-infrared autofluorescence. After a thyroid or parathyroid operation, the removed tissue is scanned with PTFinder and then checked again under normal white light. We will measure how fast (seconds) and how accurately the device finds real glands, confirmed by frozen pathology or a rapid PTH strip. About 180 adult patients at three Chinese hospitals will join. The imaging adds only a few minutes and does not change any part of the surgery. We will also record blood calcium and PTH at 1 h, 24 h, and 7 d after surgery to see whether better gland recovery lowers low-calcium risk.Collected images will also be used to train and test a deep-learning model for fully automated parathyroid recognition; model performance metrics constitute secondary outcomes.

DETAILED DESCRIPTION:
Prospective, paired, observational study at three endocrine-surgery centers. For each specimen:

PTFinder scan - stopwatch runs until the first gland is seen; all suspected glands are marked.

White-light exam - second investigator, blinded to device results, inspects the same specimen.

All marked tissue plus a random "negative" sample go to frozen section or rapid PTH strip; discrepancies are settled by permanent histology.

Outcomes

Primary - time to first gland; detection rate per specimen.

Secondary - sensitivity, specificity, PPV, NPV; post-operative PTH and calcium at 1 h, 24 h, 7 d; incidence of hypocalcaemia.

Sample size: 60 specimens per site (total = 180) gives 80 % power to detect a rise in detection rate from 70 % to 90 % (α = 0.05, McNemar).

Analysis: Paired tests for efficiency, mixed-effects models for accuracy and lab values; multiple imputation for missing data.

Safety & Oversight: PTFinder emits low-intensity NIR light only on ex-vivo tissue; no patient exposure. Device is investigational, not under an FDA IDE. Ethics approval obtained from Fujian Medical University Union Hospital IRB (FJMU-IRB-2025-PTF); other sites use the same central IRB agreement. Data are stored in a secure eCRF.

Collected images will also be used to train and test a deep-learning model for fully automated parathyroid recognition; model performance metrics constitute secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Scheduled for elective total thyroidectomy, hemithyroidectomy, or parathyroidectomy with removal of thyroid/parathyroid tissue.
* Able and willing to provide written informed consent for participation and specimen imaging.

Exclusion Criteria:

* History of neck irradiation or prior neck surgery that may distort parathyroid anatomy.
* Pregnancy or breastfeeding.
* Confirmed or suspected parathyroid carcinoma, or thyroid carcinoma requiring en-bloc parathyroid resection.
* Inability to understand the study procedures or to comply with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients undergoing thyroid or parathyroid surgery at three tertiary endocrine-surgery centers in China (Fuzhou, Xiamen, and Wenzhou). Approximately 60 participants will be enrolled per center, for a planned total of 180 surgical specimens. The cohort reflects routine clinical practice and is intended to evaluate the ex-vivo performance of the PTFinder near-infrared autofluorescence imaging device.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection Rate of Pathology-Confirmed Parathyroid Glands per Specimen (PTFinder) | Intra-operative imaging session (0-5 minutes)
  Proportion of parathyroid glands correctly located by PTFinder divided by the total number of glands confirmed on frozen section or rapid PTH strip. Unit = % (higher = better).

SECONDARY OUTCOMES:
Time to First Parathyroid Gland Identification (PTFinder) | 1 day (Same imaging session)
  Seconds from start of device scanning to first verified gland highlight (stopwatch). Lower value indicates faster localisation.
Sensitivity of PTFinder | 1 day (Same imaging session)
  True-positive glands / (true-positive + false-negative) versus frozen pathology/PTH strip. Unit = %.
Specificity of PTFinder | 1 day (Same imaging session)
  True-negative sites / (true-negative + false-positive). Unit = %.
Serum PTH Level | 1 hour , 24 hours, 7 days post-op
  Mean parathyroid hormone concentration (pg/mL) at each time-point.
Corrected Serum Calcium Level | 1 hour , 24 hours, 7 days post-op
  Mean calcium (mmol/L) adjusted for albumin.
Incidence of Hypocalcaemia | Up to 7 days post-op
  % of participants with corrected calcium <2.0 mmol/L or symptoms requiring supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, FJ, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data-NIR/RGB image files, time-to-detection, pathology confirmation, and postoperative PTH & calcium values-will be available 6 months after the primary manuscript is published, for 3 years, to qualified researchers who provide a methodologically sound proposal and sign a data-use agreement. Requests should be sent to the Principal Investigator (wangbo@fjmu.edu.cn).
Supporting Information: Study Protocol, SAP
Time Frame: "De-identified image dataset and trained AI weights will be deposited in an open repository (e.g., Zenodo) 6 months after publication, pending IRB approval."
Access Criteria: Researchers must obtain IRB approval or exemption and agree to use the data only for scientific purposes.

REFERENCES:
- [Background] Wang B, Zhou CP, Ao W, Cai SJ, Ge ZW, Wang J, Huang WY, Yu JF, Wu SB, Yan SY, Zhang LY, Wang SS, Wang ZH, Hua S, Abdelhamid Ahmed AH, Randolph GW, Zhao WX. Exploring near-infrared autofluorescence properties in parathyroid tissue: an analysis of fresh and paraffin-embedded thyroidectomy specimens. J Biomed Opt. 2025 Jan;30(Suppl 1):S13702. doi: 10.1117/1.JBO.30.S1.S13702. Epub 2024 Jul 18. PMID 39034960